CLINICAL TRIAL: NCT05127317
Title: Can Mechanical Power be Used as a Safety Precaution in Pediatric Patients?
Brief Title: Mechanical Power in Pediatric Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Ahmet YUKSEK, Asst.Prof.Dr., Bozok University
Other Study IDs: 2017-KAEK-02082021
Record Dates: First submitted 2021-11-12; First posted 2021-11-19 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Mechanical Ventilation Complication; Aediatric Anesthesia
Keywords: mechanical ventilation; pediatric anesthesia; mechanical power

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Mechanical power — In our study, mechanical power (MP) will be calculated during mechanical ventilation in patients who will be operated under general anesthesia.
  MP will be calculated with the simplified formula applied by Gattinoni et al. MPvcv: RR x Tv x (PIP-[(Pplat-PEEP)/2]) x 0.098(2) In pressure-controlled ventilation, the simplified MP formula of Becher et al. well be used.
  MPpcv: RR x Tv x (ΔPinsp + PEEP) x 0.098 (11)
  For MP calculated according to the weight of the patients; Indexed MP: MP /kg according to IBW. For the force applied to the lungs in each inspiration; Dynamic power (mJ/min): Vt x RR x [(Pplato+ tPEEP)/2]. For the driver power that provides the gas flow; Driving power (mJ/min): Vt x RR x [ (Pplat - tPEEP) / 2]. Calculating mechanical energy; Mechanical energy (mJ/kg): 0.098 x (V x kg ) x (PIP - [(P plateau- PEEP) / 2]) formulas were used

SUMMARY:
Mechanical power is the amount of energy transferred to the respiratory system of patients during each breath period. After overcoming the resistances required for respiration, the remaining energy may end up by damaging the lung parenchyma. Promising studies are showing that this amount of energy, which can be calculated mathematically, can be used as a single indicator instead of the limits used for barotrauma, volu-trauma, or atelecto-trauma in adult patients. However, the MP limit that should not be exceeded in pediatric patients is not yet clear. In this study, we present our MP calculations in pediatric anesthesia

DETAILED DESCRIPTION:
Mechanical ventilation is applied to millions of healthy and sick lungs every year in perioperative conditions and intensive care units. Meanwhile, the energy applied to the lungs by the ventilator during mechanical ventilation is usually used to overcome resistance in the chest wall and airways. Leftover energy is consumed by temperature, inflammation, and potentially lung tissue damage (1). The risk of ventilation-related damage increases in lungs with impaired homogeneity and ventilation-perfusion imbalance (1). As demonstrated by experimental and clinical studies, mechanical ventilation-induced lung injury (VILI) is associated with tidal volume, peak pressure, respiratory rate, and airflow. The physical force applied during ventilation TV increases exponentially with driving pressures (ΔPaw), flow (exponent = 2), and respiration rate (RR) (exponent = 1.4), and linearly with positive end-expiratory pressure (PEEP) (2). When the effects of these parameters are formulated, the energy applied to the lungs is revealed. This energy has been formulated as Joule/minute and has now taken its place as mechanical power (MP) in the literature. (2). A benefit of the MP calculation is that it is a single, easily calculated indicator parameter that can be used for the risks of barotrauma, volutrauma, or atelectotrauma associated with VILI. As shown in different publications, high MP values were associated with negative outcomes such as increased 30-day mortality in intensive care patients, increased length of stay in hospital and intensive care unit, and decreased number of ventilator-free days(3)(4). Cressoni et al. showed in their experimental study that MP values above 12 J/min in healthy pigs are associated with MV-related complications and this value can also be used as an alarm limit in humans(5). In addition, Costa et al found that 0.32 ± 0.14 J / min/ kg indexed MP(MP/Kg) was associated with increased mortality in ARDS patients(6). Some recent studies also support the conclusion that Mp calculation is beneficial(7)(8). For this reason, Gattinoni et al. suggests that MP limits and formula should be added to the mechanical ventilator software(2). However, studies on MP have often focused on ARDS and have been performed on intensive care patients or experimental animal models(9). Although MP is a promising safety limit with its easy computability, there are still questions about the formula and its usefulness. The success of the MP formula in perioperative situations and especially in pediatric patients has not been adequately tested. As far as we know, our study is one of the first publications to question the MP threshold in healthy pediatric cases.

In this study, our primary aim is to calculate the MP applied in pediatric cases who will undergo inguinal hernia surgery under general anesthesia.

Our other aims are the calculation of the mechanical power applied per kilogram and the other transferred energies, their comparison with the literature, and questioning the possible contribution of a mechanical power formula to safe mechanical ventilation in pediatric cases.

ELIGIBILITY:
Inclusion Criteria:

- To undergo laparoscopic lower abdomen surgery under general anesthesia under elective conditions under the age of 18

Exclusion Criteria:

- Patients in both groups weill be excluded if they had uncorrected congenital heart disease, pre-existing lung or airway disease, conditions that may decrease chest wall compliance, chronic respiratory failure requiring long-term MV, and tracheostomy.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All patients under the age of 18 who will undergo laparoscopic lower abdomen surgery under general anesthesia under elective conditions.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
median mechanical power | Measurements will be taken after half an hour of mechanical ventilation.
  mechanical force applied to the lungs during mechanical ventilation, calculated according to the formula

SECONDARY OUTCOMES:
indexed mechanical power | Data will be obtained at the beginning of the operation and after half an hour of ventilation
  mechanical power and other mechanical ventilator parameters applied according to the weight of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet YUKSEK, asst.prof, Study Chair — Yozgat Bozok Universitesi
Locations (1):
- Bozok Univesity Hospital, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kneyber MCJ. Driving Pressure and Mechanical Power: The Return of Physiology in Pediatric Mechanical Ventilation. Pediatr Crit Care Med. 2021 Oct 1;22(10):927-929. doi: 10.1097/PCC.0000000000002829. No abstract available. PMID 34605787
- [Result] Becher T, van der Staay M. Calculation of mechanical power for pressure-controlled ventilation: author's reply. Intensive Care Med. 2019 Oct;45(10):1498-1499. doi: 10.1007/s00134-019-05742-7. Epub 2019 Aug 20. No abstract available. PMID 31432217